CLINICAL TRIAL: NCT00840710
Title: Clinical Feasibility of Birth- Track II System
Acronym: BT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Barnev Ltd (Other)
Responsible Party: Clinical Trial Manager, Barnev Ltd
Other Study IDs: BT-II-IS-001
Record Dates: First submitted 2009-02-08; First posted 2009-02-10 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-02

CONDITIONS: Obstetrics; Labor
Keywords: women in active labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The Study purpose is to monitor the cervix dilation, head descent, FHR and to follow contraction in a women in active labor.

ELIGIBILITY:
Inclusion Criteria:

1. Laboring women referred to the Maternity Center in active labor (3cm dilatation and contractions).
2. Gestational age 37-42 weeks. (GA)
3. Single fetus
4. Subjects who understood, agreed and signed the informed consent form

Exclusion Criteria:

1. Women with abnormal placentation (placenta previa)
2. Abnormal fetal presentation (breech presentation)
3. Maternal History of HIV and/or blood transmitted hepatitis and/or active genital Herpes.
4. Need for immediate delivery (cord prolapsed or suspected placental abruption)

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women in active labor
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2010-02; Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, PhD, Principal Investigator — Westren Gallilie Hospital
Locations (1):
- Westren Gallilie Hospital, Nahariya, Israel